CLINICAL TRIAL: NCT01211873
Title: Safety and Efficacy Evaluation of DOTAREM® in Magnetic Resonance Imaging (MRI) in Patients With Central Nervous System (CNS) Lesions.
Brief Title: Safety and Efficacy Evaluation of DOTAREM® in MRI of Central Nervous System (CNS) Lesions
Acronym: SENTIO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: DGD-44-050
Record Dates: First submitted 2010-09-28; First posted 2010-09-30 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Diagnostic Self Evaluation; Central Nervous System Diseases
Keywords: CNS; Contrast Agent; MRI; Dotarem; Magnevist
MeSH Terms: conditions — Central Nervous System Diseases | interventions — gadoterate meglumine; Gadolinium DTPA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dotarem (gadoterate meglumine ) (Experimental): Dotarem and Magnevist were randomised as 2:1 ratio for adult patients.
  Interventions: Drug: Dotarem (gadoterate meglumine)
- Magnevist (gadopentetate dimeglumine) (Active Comparator): Dotarem and Magnevist were randomised as 2:1 ratio
  Interventions: Drug: Magnevist (gadopentetate dimeglumine)
- Dotarem 2 (gadoterate meglumine ) (Experimental): Pediatric patients were assigned to Dotarem group only.
  Interventions: Drug: Dotarem (gadoterate meglumine)

INTERVENTIONS:
Drug: Dotarem (gadoterate meglumine) — 0.1 mmol/kg by body weight, single IV injection
  Other Names: Dotarem
  Arms: Dotarem (gadoterate meglumine ); Dotarem 2 (gadoterate meglumine )
Drug: Magnevist (gadopentetate dimeglumine) — 0.1 mmol/kg by body weight, single IV injection
  Other Names: Magnevist
  Arms: Magnevist (gadopentetate dimeglumine)

SUMMARY:
The purpose of this study is to look at the safety (what are the side effects)and efficacy (how well does it work) of Dotarem® when used in taking images of the brain / spine. The results will be compared to the results of MRI taken without Dotarem.

DETAILED DESCRIPTION:
This is a study involving the use of Magnetic Resonance Imaging (MRI) contrast agents called Dotarem®. The purpose of this study is to look at the safety (what are the side effects) and efficacy (how well does it work) of Dotarem® when used for taking images of the brain and spine. The results of the MRI will be compared to the results of images taken without Dotarem®.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject and pediatric subjects (aged greater than or equal to two (2) years).
* Is referred for a contrast-enhanced MRI of the CNS based on the results of a previous imaging procedure.
* Female of childbearing potential patients must have effective contraception (contraceptive pill or intra-uterine device) or be surgically sterilized or post-menopausal (minimum 12 months amenorrhea), or have a documented negative urine pregnancy test within 24 hours prior to study MRI.
* Has been fully informed about the study, and has consented to participate.

Exclusion Criteria:

* Having acute or chronic grade IV or V renal insufficiency.
* Known class III/IV congestive heart failure.
* Suffering from long QT syndrome.
* Unstable health condition or circumstances (e.g. suffering from severe claustrophobia).
* Having any contraindications to MRI such as a pace-maker, magnetic material or any other conditions that would preclude proximity to a strong magnetic field.
* Known allergy to Gadolinium chelates.
* Having received any contrast agent within 3 days prior to study contrast administration, or is scheduled to receive any contrast agent within 24 hours after the study contrast administration.
* Pregnant, breast feeding, or planning to become pregnant during the trial.
* Previously participated in this trial.
* Having participated within 30 days in another clinical trial involving an investigational drug.
* Any condition which, based on the investigator's clinical judgement, would prevent the patient from completing all trial assessments and visits.
* Inability or unwillingness to cooperate with the requirements of this trial.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Maravilla, MD, Principal Investigator — University of Wasington School of Medicine
Locations (52):
- United States (20):
  - University of Alabama at Birmingham, UABMC, Birmingham, Alabama
  - University Medical Center, Tucson, Arizona
  - University medical center, Tucson, Arizona
  - Desert Medical Imaging, Indian Wells, California
  - Sunrise Clinical Research, Inc., Hollywood, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Precise Clinical Research Solutions, Topeka, Kansas
  - University of Louisville Hospital, Louisville, Kentucky
  - Neurocare Center for Research, Brookline, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - QUEST Research Institute, Farmington Hills, Michigan
  - Gruss Magnetic resonance Research Clinic, New York, New York
  - WestImage - Division of Research, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas - Health Science Center, San Antonio, Texas
  - UTHSCSA, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Argentina (3):
  - Centro de Diagnóstico, Buenos Aires
  - Hospital Italiano, Buenos Aires
  - TCBA, Buenos Aires
- Austria (3):
  - Univ.-institut f.Radiodiagnostik, Salzburg
  - Landesklinikum Tulln, Tulln
  - Medical University of Vienna, Vienna
- Brazil (2):
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
  - Universidade Federal de São Paulo / UNIFESP, São Paulo
- Chile (2):
  - Departamento de Neuroradiologia, Santiago
  - Instituto de Neurocirugia Dr. Asenjo,, Santiago
- France (6):
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Roger Salengro- CRHU de Lille, Lille
  - Hôpital Gui De Chauliac, Montpellier
  - Centre Hospitalier Sainte Anne, Paris
  - Radiologie A - Hôpital de la Milétrie, Poitiers
  - Fédération d'Imagerie Médicale,Hôpital Pontchaillou, Rennes
- Germany (7):
  - University Hospital Charite, Berlin
  - Krankenhaus Nordwest GmbH, Frankfurt
  - University Hospital Frankfurt, Frankfurt am Main
  - University of Heidelberg, Heidelberg
  - University of Leipzig, Leipzig
  - University Hospital Mannheim, Mannheim
  - University Hospital LMU Munich, Munich
- Italy (3):
  - Istituto di Radiologia, Florence
  - Neuroradiologia,II Università Di Napoli, Napoli
  - Azienda Ospedaliera S. Andrea, Roma
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Seoul National Unversity Hospital, Seoul
- Spain (3):
  - Hospital Vall d´Hebron, Barcelona
  - Hospital Clinico Universitario San Carlos, Madrid
  - Complejo Hospitalario Universitario de Vigo - Serviço de radiologia, Vigo
- University Department of Radiology, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient First Visit : 16 Sept 2010 Last patient Last Visit : 16 Nov 2011 Locations: radiology departments
Pre-assignment Details: Any patient who did not fulfill eligibility criteria was not randomized / assigned to a treatment group.
Groups:
- Dotarem (Gadoterate Meglumine): Dotarem and Magnevist were randomised as 2:1 ratio for adult patients.
- Dotarem 2 (Gadoterate Meglumine): Pediatric patients were assigned to Dotarem group only
Period: Overall Study
Arm/Group | Dotarem (Gadoterate Meglumine) | Magnevist (Gadopentetate Dimeglumine) | Dotarem 2 (Gadoterate Meglumine)
Started | 245 | 119 | 38
Completed | 240 | 117 | 36
Not Completed | 5 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Magnevist (Gadopentetate Dimeglumine): adults received Magnevist as 1:2 ratio compared to Dotarem
- Dotarem (Gadoterate Meglumine): adults received Dotarem as 2:1 ratio compared to Magnevist.
- Dotarem 2 (Gadoterate Meglumine): All children were assigned to Dotarem
- Total: Total of all reporting groups
Arm/Group | Magnevist (Gadopentetate Dimeglumine) | Dotarem (Gadoterate Meglumine) | Dotarem 2 (Gadoterate Meglumine) | Total
Number analyzed (Participants) | 119 | 245 | 38 | 402
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 38 | 38
  Between 18 and 65 years | 89 | 185 | 0 | 274
  >=65 years | 30 | 60 | 0 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.95 (14.43) | 53.17 (14.35) | 9.29 (4.49) | 49.8 (19.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 131 | 22 | 218
  Male | 54 | 114 | 16 | 184
Region of Enrollment [Number; unit: participants]
  United States | 30 | 65 | 17 | 112
  France | 13 | 30 | 0 | 43
  Argentina | 12 | 22 | 14 | 48
  Brazil | 5 | 8 | 4 | 17
  Spain | 2 | 8 | 0 | 10
  Austria | 10 | 20 | 0 | 30
  Chile | 3 | 5 | 3 | 11
  Germany | 20 | 40 | 0 | 60
  United Kingdom | 3 | 6 | 0 | 9
  Italy | 7 | 15 | 0 | 22
  Korea, Republic of | 14 | 26 | 0 | 40

OUTCOME MEASURES:

1. Primary Outcome: MRI Lesion Visualization (Border Delineation, Internal Morphology and Contrast Enhancement) at Patient Level for Both "Pre" and "Paired" Evaluation
Description: To demonstrate the superiority of combined unenhanced and Dotarem enhanced MRI (PAIRED) compared to unenhanced MRI (PRE) in terms of lesion visualization.
  Unenhanced MRI refers to MRI before administration of contrast agent. Enhanced MRI refers to MRI after contrast agent injection. "Pre" refers to unenhanced MRI. "PAIRED" refer to combined unenhanced and enhanced MRI.
  The measure used a specific scale with 3-point levels to assess lesion visualization. At lesion level, the scale range is from 0 through 1 to 2. Score 0 means a worse outcome and score 2 means a better outcome. Patient score is the sum of all lesion scores. Up to 5 of the largest representative lesions were assessed. At patient level, the maximum score is 10, minimum score is 0.
Time Frame: up to 24 hours
Population: The primary analysis was performed at the patient level using off-site readings by 3 readers. The number of participants for analysis depended on the number of evaluable cases (PRE and PAIRED) determined by each reader. Only adult participants were included in this data set.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Dotarem (Gadoterate Meglumine) - PRE: Any sequence acquired prior to injection of Dotarem was pooled as PRE
- Dotarem (Gadoterate Meglumine) - PAIRED: All sequences pre- and post-injection of Dotarem were pooled as PAIRED
Arm/Group | Dotarem (Gadoterate Meglumine) - PRE | Dotarem (Gadoterate Meglumine) - PAIRED
Number analyzed (Participants) | 224 | 235
units on a scale
  Border Delineation Blinded Reader 1 | 1.06 (1.23) | 3.30 (2.64)
  Border Delineation Blinded Reader 2 | 1.62 (1.43) | 4.49 (2.94)
  Border Delineation Blinded Reader 3 | 1.43 (1.29) | 2.54 (2.30)
  Internal Morphology Blinded Reader 1 | 0.97 (1.05) | 3.70 (2.63)
  Internal Morphology Blinded Reader 2 | 1.76 (1.24) | 4.49 (2.93)
  Internal Morphology Blinded Reader 3 | 1.45 (1.13) | 2.93 (2.30)
  Contrast Enhancement Blinded Reader 1 | 0.01 (0.20) | 3.11 (2.52)
  Contrast Enhancement Blinded Reader 2 | 0.01 (0.15) | 3.73 (2.67)
  Contrast Enhancement Blinded Reader 3 | 0.01 (0.13) | 2.95 (2.44)
Statistical Analysis 1: Comparison: Dotarem (Gadoterate Meglumine) - PRE vs Dotarem (Gadoterate Meglumine) - PAIRED; Test type: Superiority; p < 0.001, Regression, Logistic

2. Secondary Outcome: Image Quality Score
Description: Image quality was evaluated for each lesion according to a 3-point scale with the following grades; poor (1), fair (2) or good (3), and an overall score per patient was calculated. At patient level, the maximum score is 3, minimum score is 1. Higher scores mean a better image quality.
Time Frame: up to 24 hours
Population: The number of participants for analysis depended on the number of evaluable cases (PRE and PAIRED) determined by each reader. Only adult participants are included in this data set.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Magnevist (Gadopentetate Dimeglumine) - PRE: Any sequence acquired prior to injection of Magnevist was pooled as PRE
- Magnevist (Gadopentetate Dimeglumine) - PAIRED: All sequences pre- and post-injection of Magnevist were pooled as PAIRED
Arm/Group | Dotarem (Gadoterate Meglumine) - PRE | Dotarem (Gadoterate Meglumine) - PAIRED | Magnevist (Gadopentetate Dimeglumine) - PRE | Magnevist (Gadopentetate Dimeglumine) - PAIRED
Number analyzed (Participants) | 224 | 235 | 113 | 116
units on a scale
  Reader 1: number analyzed (Participants) | 224 | 230 | 111 | 114
  Reader 1 | 1.41 (0.52) | 2.98 (0.20) | 1.42 (0.53) | 2.96 (0.26)
  Reader 2: number analyzed (Participants) | 224 | 230 | 113 | 114
  Reader 2 | 1.72 (0.45) | 3.00 (0) | 1.74 (0.44) | 2.98 (0.19)
  Reader 3: number analyzed (Participants) | 222 | 235 | 113 | 116
  Reader 3 | 2.00 (0.07) | 2.99 (0.11) | 1.99 (0.09) | 2.99 (0.09)
Statistical Analysis 1: Comparison: Dotarem (Gadoterate Meglumine) - PRE vs Dotarem (Gadoterate Meglumine) - PAIRED; Test type: Superiority; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: Magnevist (Gadopentetate Dimeglumine) - PRE vs Magnevist (Gadopentetate Dimeglumine) - PAIRED; Test type: Superiority; p < 0.001, Regression, Logistic

3. Secondary Outcome: Diagnostic Confidence Score
Description: Level of diagnostic confidence when evaluating the MRI modalities was graded using a 5-point scale as nil (1), poor (2), moderate (3), high (4) and excellent (5).
Time Frame: up to 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dotarem (Gadoterate Meglumine) - PRE | Dotarem (Gadoterate Meglumine) - PAIRED | Magnevist (Gadopentetate Dimeglumine) - PRE | Magnevist (Gadopentetate Dimeglumine) - PAIRED
Number analyzed (Participants) | 224 | 235 | 113 | 116
units on a scale
  Reader 1 | 3.04 (0.90) | 4.59 (0.64) | 3.11 (0.86) | 4.66 (0.64)
  Reader 2 | 2.84 (0.61) | 4.89 (0.31) | 2.85 (0.59) | 4.92 (0.36)
  Reader 3 | 3.47 (1.22) | 4.41 (0.98) | 3.59 (1.29) | 4.59 (0.81)
Statistical Analysis 1: Comparison: Dotarem (Gadoterate Meglumine) - PRE vs Dotarem (Gadoterate Meglumine) - PAIRED; Test type: Superiority; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: Magnevist (Gadopentetate Dimeglumine) - PRE vs Magnevist (Gadopentetate Dimeglumine) - PAIRED; Test type: Superiority; p < 0.001, Regression, Logistic

4. Secondary Outcome: Number of Lesions
Description: The number of lesions for which observations could be made was calculated for each MRI modality and results are summarized per patient
Time Frame: up to 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of lesions
Arm/Group | Dotarem (Gadoterate Meglumine) - PRE | Dotarem (Gadoterate Meglumine) - PAIRED | Magnevist (Gadopentetate Dimeglumine) - PRE | Magnevist (Gadopentetate Dimeglumine) - PAIRED
Number analyzed (Participants) | 224 | 235 | 113 | 116
Number of lesions
  Reader 1 | 1.97 (3.16) | 2.69 (4.71) | 1.98 (3.85) | 4.19 (10.54)
  Reader 2 | 2.29 (3.69) | 3.16 (5.21) | 2.60 (5.42) | 4.50 (9.95)
  Reader 3 | 1.97 (2.99) | 2.46 (4.53) | 2.15 (3.97) | 3.97 (10.02)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from patient consent signature to the end of the last visits, maximum duration is 29 days.
Description: Participants at risk were subjects exposed to contrast agent administration. In Dotarem group, 240 adults were injected, Dotarem group 2, 38 children were injected (2 children were withdrawn after agent administration) and in Magnevist group, 117 adults were injected.
Groups:
- Dotarem (Gadoterate Meglumine ): Dotarem and Magnevist were randomised as 2:1 ratio for adults
- Dotarem 2 (Gadoterate Meglumine ): children were only assigned to Dotarem
Arm/Group | Dotarem (Gadoterate Meglumine ) | Magnevist (Gadopentetate Dimeglumine) | Dotarem 2 (Gadoterate Meglumine )
All-Cause Mortality (participants affected / at risk) | 0/240 | 0/117 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/240 | 1/117 | 1/38
Other Adverse Events (participants affected / at risk) | 12/240 | 9/117 | 8/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem (Gadoterate Meglumine ) (N=240) | Magnevist (Gadopentetate Dimeglumine) (N=117) | Dotarem 2 (Gadoterate Meglumine ) (N=38)
small intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — not related
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — not related
neurological decompensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — not related
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dotarem (Gadoterate Meglumine ) (N=240) | Magnevist (Gadopentetate Dimeglumine) (N=117) | Dotarem 2 (Gadoterate Meglumine ) (N=38)
injection site pain (General disorders) | 3 | 1 | 0
injection site hematoma (General disorders) | 0 | 3 | 0
extravasation (General disorders) | 1 | 2 | 0
chest pain (General disorders) | 0 | 2 | 0
blood urine present (Investigations) | 2 | 0 | 1
nausea (Gastrointestinal disorders) | 3 | 0 | 1
headache (Nervous system disorders) | 1 | 1 | 2
dizziness (Nervous system disorders) | 1 | 0 | 1
vomiting (Gastrointestinal disorders) | 1 | 0 | 1
asthenia (General disorders) | 0 | 0 | 1
application site erythema (General disorders) | 0 | 0 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished data given to the investigator may be transmitted to a third party without prior approval of the sponsor in writing. The data are the exclusive property of Guerbet.

The investigator undertakes to submit to Guerbet any draft articles or papers related to this study within 30 days of their submission to the scientific review or the congress scientific committee.

All written or oral papers and publications must have the joint agreement of the investigator and the sponsor.